CLINICAL TRIAL: NCT05783466
Title: Bioactive Dairy Lipids to Manage Cardiometabolic Risk in Obesity
Brief Title: Dairy Lipids and Cardiometabolic Risk
Acronym: DAILICATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Laboratoire de Recherche en Cardiovasculaire, Métabolisme, Diabétologie et Nutrition (Unknown); Centre de Recherche en Nutrition Humaine Rhone-Alpe (Other); Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL22_0461; 2022-A02415-38 (Other: ID-RCB)
Record Dates: First submitted 2023-02-16; First posted 2023-03-24 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Morbid Obesity
Keywords: Obesity; Nutrition; Dietary intervention; Weight loss; Metabolism; Dairy; Fat; Milk polar lipids
MeSH Terms: conditions — Obesity, Morbid; Obesity; Weight Loss; Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low-fat dairy products within a dietary handling for weight loss (Other): 3 servings/day of low-fat dairy products: 1 serving of low-fat cheese, 1 serving of low-fat yogurt and 1 serving of (semi-)skimmed milk.
  Interventions: Other: Low-fat dairy products
- Whole-fat dairy products within a dietary handling for weight loss (Experimental): 3 servings/day of whole-fat dairy products: 1 serving of whole cheese, 1 serving of whole yogurt and 1 serving of whole milk.
  Interventions: Other: Whole-fat dairy products
- Whole-fat dairy products enriched with milk polar lipids within a dietary handling for weight loss (Experimental): 3 servings/day of whole-fat dairy products (1 milk, 1 yogurt, 1 cheese) among which 1 serving/day is enriched with milk polar lipids via butterier.
  Interventions: Other: Milk polar lipid enriched whole-fat dairy products

INTERVENTIONS:
Other: Low-fat dairy products — 3-month intervention
  Arms: Low-fat dairy products within a dietary handling for weight loss
Other: Whole-fat dairy products — 3-month intervention
  Arms: Whole-fat dairy products within a dietary handling for weight loss
Other: Milk polar lipid enriched whole-fat dairy products — 3-month intervention
  Arms: Whole-fat dairy products enriched with milk polar lipids within a dietary handling for weight loss

SUMMARY:
It is a randomized parallel arm intervention study in adults with severe obesity. The objective is to demonstrate that within a dietary handling for weight loss, the daily ingestion during 3 months of whole dairy products enriched with milk polar lipids or whole dairy products decreases to a greater extent fasting plasma apolipoprotein B concentrations than the daily ingestion of low-fat dairy products (control group).

Metabolic parameters will be assessed before and after the 3-month intervention, both at fasting and in postprandial period after the consumption of standardized meals.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18-70 years
* Body Mass Index (BMI) between 35 and 60 kg/m2 inclusive
* Stable body weight (weight change +/- 5 % for 3 months prior to screening)
* Consumption of at least 1 serving/day of dairy products made from cow's milk
* Informed consent

Exclusion Criteria:

* History of bariatric or digestive surgery or disease interfering with main outcomes
* Drinking more than 3 glasses of alcohol per day (>30g/day)
* Pregnancy, parturiency or breastfeeding
* Food allergies or intolerance to dairy products
* Dietary restriction (vegetarian or lactovegetarian) or high protein diet
* Use of dietary supplements
* Treated with lipid lowering drugs (fibrates, statins, anti-PCSK9, ezetimibe, cholestyramine) within the last 6 weeks before study entry
* Treated with insulin, GLP-1 analogs, acarbose, corticoids, beta-blockers.
* Medications interfering with intestinal microbiota (beta-lactamines within 3 months before the study or laxatives)
* Smoking ≥ 5 cigarettes/day during the past 6 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Total plasma apolipoprotein B concentration | day 0 and day 90
  Change in fasting total plasma apolipoprotein B concentration after 3-month intervention, measured by ELISA.

SECONDARY OUTCOMES:
Changes in weight | day 0 and day 90
  Changes in weight after 3-month intervention.
Anthropometric measurements 2 | day 0 and day 90
  Changes in waist and hip circumferences after 3-month intervention.
Body mass composition measurements | day 0 and day 90
  Change in body mass composition (lean mass, fat mass) after 3-month intervention, analyzed by impedancemeter
Plasma lipid concentrations after 3-month intervention, measured using standard laboratory methods | day 0 and day 90 for fasting and postprandial measurements. • For postprandial measurements: times 60 minutes-120 minutes -180 minutes -240 minutes -270 minutes -300 minutes -360 minutes
  Changes in plasma concentrations of triglycerides
Plasma lipid concentrations after 3-month intervention, measured using standard laboratory methods 2 | day 0 and day 90 for fasting and postprandial measurements. For postprandial measurements: times 120 minutes -180 minutes -240 minutes -270 minutes -300 minutes.
  Changes in plasma concentrations of total cholesterol
Plasma lipid concentrations after 3-month intervention, measured using standard laboratory methods 3 | day 0 and day 90 for fasting and postprandial measurements. For postprandial measurements: time 360 minutes.
  Changes in plasma concentrations of LDL-cholesterol
Plasma lipid concentrations after 3-month intervention, measured using standard laboratory methods 4 | day 0 and day 90 for fasting and postprandial measurements. For postprandial measurements: time 360 minutes.
  Changes in plasma concentrations of HDL-cholesterol
Plasma lipid concentrations after 3-month intervention, measured using standard laboratory methods 5 | day 0 and day 90 for fasting and postprandial measurements. For postprandial measurements: times 120 minutes -240 minutes -300 minutes.
  Changes in plasma concentrations of apoB100
Plasma lipid concentrations after 3-month intervention, measured using standard laboratory methods 6 | day 0 and day 90 for fasting and postprandial measurements. For postprandial measurements: times 120 minutes -240 minutes -300 minutes - 360 minutes
  Changes in plasma concentrations of apoB48
Plasma lipid concentrations after 3-month intervention, measured using standard laboratory methods 7 | day 0 and day 90 for fasting and postprandial measurements. For postprandial measurements:times 360 minutes.
  Changes in plasma concentrations of apoA1
Plasma lipid concentrations after 3-month intervention, measured using standard laboratory methods 8 | day 0 and day 90 for fasting and postprandial measurements. For postprandial measurements: times 120 minutes -240 minutes
  Changes in plasma concentrations of unesterified fatty acids
Glucose concentrations after 3-month intervention, measured using standard laboratory methods | day 0 and day 90 for fasting and postprandial measurements. For postprandial measurements: times 120 minutes -240 minutes
  Changes in plasma concentrations of glucose
Glucose concentrations after 3-month intervention, measured using standard laboratory methods 2 | day 0 and day 90 for fasting and postprandial measurements. For postprandial measurements: times 120 minutes -240 minutes
  Changes in plasma concentrations of insulin
Targeted plasma lipidomics after 3-month intervention | day 0 and day 90 for fasting and postprandial measurements For postprandial measurements :times 120 minutes -240 minutes -300 minutes -360 minutes.
  Changes in plasma concentrations of phospholipids
Targeted plasma lipidomics after 3-month intervention 2 | day 0 and day 90 for fasting and postprandial measurements For postprandial measurements :times 120 minutes -240 minutes -300 minutes -360 minutes.
  Changes in plasma concentrations of sphingolipids (sphingomyelins and ceramides)
Targeted plasma lipidomics after 3-month intervention 3 | day 0 and day 90 for fasting and postprandial measurements For postprandial measurements :times 120 minutes -240 minutes -300 minutes -360 minutes.
  Changes in plasma concentrations of lysophospholipids
Targeted plasma lipidomics after 3-month intervention 4 | day 0 and day 90 for fasting and postprandial measurements For postprandial measurements :times 120 minutes -240 minutes -300 minutes -360 minutes.
  Changes in plasma concentrations of fatty acids in plasma total lipids
Targeted plasma lipidomics after 3-month intervention 5 | day 0 and day 90 for fasting and postprandial measurements For postprandial measurements :times 120 minutes -240 minutes -300 minutes -360 minutes.
  Changes in plasma concentrations of phospholipids
Targeted chylomicrons of plasma after 3-month intervention | day 0 and day 90 for fasting and postprandial measurements For postprandial measurements :times 120 minutes -240 minutes -300 minutes -360 minutes.
  Changes in concentrations of triglycerides
Targeted chylomicrons of plasma after 3-month intervention 2 | day 0 and day 90 for fasting and postprandial measurements For postprandial measurements :times 120 minutes -240 minutes -300 minutes -360 minutes.
  Changes in concentrations of cholesterol
Targeted chylomicrons of plasma after 3-month intervention 3 | day 0 and day 90 for fasting and postprandial measurements For postprandial measurements :times 120 minutes -240 minutes -300 minutes -360 minutes.
  Changes in concentrations of sphingolipids
Targeted chylomicrons of plasma after 3-month intervention 4 | day 0 and day 90 for fasting and postprandial measurements For postprandial measurements :times 120 minutes -240 minutes -300 minutes -360 minutes.
  Changes in concentrations of fatty acids
Inflammation markers | day 0 and day 90 for fasting and postprandial measurements.
  Changes in adiponectin
Inflammation markers 2 | day 0 and day 90 for fasting and postprandial measurements.
  Changes in CRP
Inflammation markers 3 | day 0 and day 90 for fasting and postprandial measurements.
  Changes in cytokines
Inflammation markers 4 | day 0 and day 90 for fasting and postprandial measurements.
  Changes in LBP
Inflammation markers 5 | day 0 and day 90 for fasting and postprandial measurements.
  Changes in endotoxins
Inflammation markers 6 | day 0 and day 90 for fasting and postprandial measurements.
  Changes in CD14
Inflammation markers 7 | day 0 and day 90 for fasting and postprandial measurements.
  Gene expressions of inflammation markers after 3-month intervention, measured with dedicated kits and PAXgene kit
Platelet activation markers | day 0 and day 90 for fasting and postprandial measurements. For postprandial measurements,times 120 minutes-240 minutes-300 minutes -360 minutes.
  Changes in thromboxane B2 concentrations in platelets (from blood donors) stimulated by lipoproteins (chylomicrons and HDL) after 3-month intervention, measured with an ELISA kit.
  Differences in the percents of aggregation of platelets incubated with lipoproteins (chylomicrons and HDL) after 3-month intervention, assessed by light transmission aggregometry.
Oxidative stress marker | day 0 and day 90
  Changes in urinary concentrations of 8-iso-PGF2 alpha isoprostane after 3-month intervention, determined with an ELISA kit
Markers of immune cells | day 0 and day 90
  PBMC
Markers of immune cells 2 | day 0 and day 90
  Complete blood counts
Intestinal microbiota after 3-month intervention. | day 0 and day 90
  Changes in microbiome composition and diversity (alpha, beta) of feces (16S analysis)
Intestinal microbiota after 3-month intervention 2 | day 0 and day 90
  Changes in fecal concentrations of microbiota-derived metabolites (coprostanol, short chain fatty acids (SCFA), calprotectin)
Questionnaires on physical activity | day 0 and day 90
  International Physical Activity Questionnaire ([i] ëinactive, [ii] ëminimally active, [iii] ëHEPA activeí (health enhancing physical activity; a high active category).)
Questionnaires on digestive comfort | day 0 and day 90
  Liker scale
Questionnaires on digestive comfort | day 0 and day 90
  Bristol stool scale
Questionnaires on product satiety | day 0 and day 90
  Satiety from visual analog scale (VAS)
Questionnaires food intake | day 0 and day 90
  Three-factor eating questionnaire (TFEQ)
Questionnaires on product appreciation | day 0 and day 90
  Product appreciation questionnaire
Dietary intake questionnaire | day 0 and day 90
  Dietary record questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre de Recherche en Nutrition Humaine Rhône-Alpes, Pierre-Bénite
  - Centres Hospitalier Lyon Sud, Service d'Endocrinologie-Diabète-Nutrition, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No